CLINICAL TRIAL: NCT05346042
Title: Safe and Timely Cessation of Isolation of Patients With COVID-19, The SCIP-COVID-19
Brief Title: Safe and Timely Cessation of Isolation of Patients With COVID-19 (The SCIP-COVID-19) Study
Acronym: SCIP-COVID19
Status: Active, not recruiting | Type: Observational
Sponsor: Anne Voor in 't holt (Other)
Collaborators: Maasstad Hospital (Other); Medisch Spectrum Twente (Other); Elisabeth-TweeSteden Ziekenhuis (Other); Julius Center (Other); HagaZiekenhuis (Other); Leiden University Medical Center (Other); Radboud University Medical Center (Other)
Responsible Party: Sponsor-Investigator, Anne Voor in 't holt, Epidemiologist, Assistant Professor, Erasmus Medical Center
Organization: Erasmus Medical Center (Other)
Other Study IDs: 113189; 10430102110003 (Other Grant/Funding Number: ZonMw)
Record Dates: First submitted 2022-04-25; First posted 2022-04-26 (Actual); Last update posted 2025-03-05 (Actual); Status verified 2025-03

CONDITIONS: COVID-19
Keywords: COVID-19; infectiousness duration; isolation; infection prevention control measures
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — serum surplus material (samples with DNA) + Stored (frozen) longitudinal nasopharyngeal swabs (samples without DNA)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Confirmed Covid-19: All adult COVID-19 patients and health care workers tested positive in the 7 participating hospitals identified between the end of February 2020 and December 2021.
  Interventions: Other: duration infectiousness

INTERVENTIONS:
Other: duration infectiousness — is the probability and the duration of being infectious in hospitalized COVID-19 patients, consequently influencing the decision on cessation of isolation

SUMMARY:
Rationale:

In the treatment, care and isolation of COVID-19 patients, one of the most important issues is determining the duration of infectiousness. The current Dutch guideline advises at least 14 days of isolation for seriously ill patients, which is the case for most admitted patients, and at least 21 days for intubated patients. It is believed that in most cases this isolation duration is too long, which is highly undesirable for patients staying in closed single-occupancy rooms. This is known to result in limited contact with healthcare workers (HCW) and to be associated with a higher level of depression among patients. The longer the isolation, the higher the workload for HCW and the higher the costs (e.g. with about 0.5 million admission days in the Netherlands, these work out at about €14 million on personal protective equipment [PPE] and cleaning alone). Additionally, isolation demands a larger healthcare workforce, yielding less capacity to provide other care to non-COVID-19 patients, with numerous other consequences. On the other hand, it is possible that some patients were discontinued from isolation too early, leading to a risk of transmission to other patients and to HCW. In conclusion, duration of isolation should be as short as possible for proper patient flow and to avoid unnecessary burden to patients and HCW, and thus to healthcare in general. Therefore, there is an urgent need to define the period of infectiousness of COVID-19. We will develop a safe and effective algorithm for decision on timely discontinuation of isolation of COVID-19 hospitalized patients.

Objective:

The ultimate goal of this project is to produce new evidence-based criteria for the termination of isolation of hospitalized COVID-19 patients that are safe (very low subsequent risk of transmission to other patients or healthcare workers) while reducing the number of unnecessary days in isolation (thereby improving quality of life of patients, reducing hospital costs, and making optimal use of the scarce number of isolation beds). Multiple sources of data and evidence will be integrated to arrive at these new criteria.

DETAILED DESCRIPTION:
Rationale:

In the treatment, care and isolation of COVID-19 patients, one of the most important issues is determining the duration of infectiousness. The current Dutch guideline advises at least 14 days of isolation for seriously ill patients, which is the case for most admitted patients, and at least 21 days for intubated patients. It is believed that in most cases this isolation duration is too long, which is highly undesirable for patients staying in closed single-occupancy rooms. This is known to result in limited contact with healthcare workers (HCW) and to be associated with a higher level of depression among patients. The longer the isolation, the higher the workload for HCW and the higher the costs (e.g. with about 0.5 million admission days in the Netherlands, these work out at about €14 million on personal protective equipment [PPE] and cleaning alone). Additionally, isolation demands a larger healthcare workforce, yielding less capacity to provide other care to non-COVID-19 patients, with numerous other consequences. On the other hand, it is possible that some patients were discontinued from isolation too early, leading to a risk of transmission to other patients and to HCW. In conclusion, duration of isolation should be as short as possible for proper patient flow and to avoid unnecessary burden to patients and HCW, and thus to healthcare in general. Therefore, there is an urgent need to define the period of infectiousness of COVID-19. We will develop a safe and effective algorithm for decision on timely discontinuation of isolation of COVID-19 hospitalized patients.

Objective:

The ultimate goal of this project is to produce new evidence-based criteria for the termination of isolation of hospitalized COVID-19 patients that are safe (very low subsequent risk of transmission to other patients or healthcare workers) while reducing the number of unnecessary days in isolation (thereby improving quality of life of patients, reducing hospital costs, and making optimal use of the scarce number of isolation beds). Multiple sources of data and evidence will be integrated to arrive at these new criteria.

Study design:

This is a retrospective cohort and technical laboratory study.

Study population:

All adult COVID-19 patients tested positive in the 7 participating hospitals identified between the end of February 2020 and December 2021.

Main study endpoint:

The main outcome of interest is the probability and the duration of being infectious in hospitalized COVID-19 patients, consequently influencing the decision on cessation of isolation.

ELIGIBILITY:
Inclusion Criteria:

In order to be eligible to participate in this study, a subject must meet all of the following criteria:

* Admission for COVID-19 and tested positive between the end of February 2020 and December 1st 2021.
* Admission for other reasons than COVID-19, but during hospital stay detected with COVID-19.
* Patients ≥18 years old.

Exclusion Criteria:

A potential subject who meets any of the following criteria will be excluded:

* Adult patients with registered opt-out for using clinical and/or laboratory data.
* Patients <18 years old.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All adult COVID-19 patients tested positive in the 7 participating hospitals between the end of February 2020 and December 2021.
Sampling Method: Probability Sample
Enrollment: 7000 (Estimated)
Dates: Start 2022-12-01 (Actual); Primary Completion 2025-02-01 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
the probability and the duration of being infectious in hospitalized COVID-19 patients, consequently influencing the decision on cessation of isolation | Between the end of February 2020 and December 2021
  the probability and the duration of being infectious in hospitalized COVID-19 patients, consequently influencing the decision on cessation of isolation

SECONDARY OUTCOMES:
Quantitative Ct-value of RT-PCR | Between the end of February 2020 and December 2021
  The quantitative Ct-value of RT-PCR as reference standard
Quantitative SARS-CoV-2 N-Ag concentration in pg/mL | Between the end of February 2020 and December 2021
  The quantitative SARS-CoV-2 N-Ag concentration in pg/mL
Qualitative rapid Ag-test | Between the end of February 2020 and December 2021
  The rapid Ag-test in qualitative form

CONTACTS AND LOCATIONS:
Overall Officials: Margreet C Vos, Prof. dr., Principal Investigator — Erasmus Medical Center
Locations (1):
- Erasmus Medical Center, Rotterdam, South Holland, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
Other researchers will be able to find the metadata in the data repository on the COVID-19 national Health-RI portal. They could express their interest in the dataset through a.voorintholt@erasmusmc.nl. After meeting the sharing and reuse conditions and approval of the PI, data access will be provided through the COVID-19 national health RI portal.
Supporting Information: Study Protocol, SAP
Time Frame: At least 10 years
Access Criteria: Researchers could express their interest in the dataset through a.voorintholt@erasmusmc.nl. After meeting the sharing and reuse conditions and approval of the PI, data access will be provided through the COVID-19 national health RI portal.